CLINICAL TRIAL: NCT01161381
Title: Evaluation Of Patients With Suspected Obstructive Sleep Apnea - Hypopnea Syndrome Using Two Models Based on Nonlinear Analysis Of Respiratory Signals
Brief Title: Evaluation Of Patients With Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) Based on Nonlinear Analysis Of Respiratory Signals
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Greek State Scholarship Foundation (Unknown)
Responsible Party: Lab of Medical Informatics, Aristotle University of Thessaloniki
Other Study IDs: EK1001
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2005-12

CONDITIONS: Obstructive Sleep Apnea Syndrome (OSAS)
Keywords: OSAHS; nonlinear analysis; polysomnography; biosignal analysis; DFA; APEN; LLE
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Subjects that underwent night polysomnography with an observed Apnea-Hypopnea Index (AHI) < 5.
  Interventions: Device: Estimation of nonlinear indices from Polysomnography
- OSAHS patients: Subjects that underwent night polysomnography with an observed Apnea-Hypopnea Index (AHI) > 5.
  Interventions: Device: Estimation of nonlinear indices from Polysomnography

INTERVENTIONS:
Device: Estimation of nonlinear indices from Polysomnography — All subjects underwent full night polysomnography. Three nonlinear indices (Largest Lyapunov Exponent, Detrended Fluctuation Analysis and Approximate Entropy) were extracted from three biosignals (airflow from a nasal cannula, thoracic movement and Oxygen saturation) providing input to a data mining application for the creation of predictive models for AHI.
  Other Names: polysomnography device: Somnologica 7000, Flaga; Iceland

SUMMARY:
Objective: Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) is a common sleep disorder requiring the time and money consuming full polysomnography to be diagnosed. Alternative methods for initial evaluation are sought. The investigators aim was the prediction of Apnea-Hypopnea Index (AHI) in patients suspected to suffer from OSAHS using two models based on nonlinear analysis of three biosignals during sleep.

Methods: One hundred patients referred to a Sleep Unit underwent full polysomnography. Three nonlinear indices (Largest Lyapunov Exponent, Detrended Fluctuation Analysis and Approximate Entropy) were extracted from three biosignals (airflow from a nasal cannula, thoracic movement and Oxygen saturation) providing input to a data mining application for the creation of predictive models for AHI.

DETAILED DESCRIPTION:
Patients referred to the Sleep Unit of a tertiary hospital in northern Greece during the years 2005-2008 and who accepted to sign the informed consent form were included in the study. One out of every five consecutive patients was selected in order to ensure randomization. The study protocol was approved by the ethics committee of the hospital. All the subjects reported symptoms consistent with OSAHS and had no significant comorbidities. The presence of dementia, neuromuscular disorders, overlap syndrome or severe cardiac problems was an exclusion criterion for the participants. The subjects underwent full overnight attended polysomnography (Somnologica 7000, Flaga; Iceland) according to standard criteria including respiratory recordings of thoracic and abdominal movements, nasal flow by pressure cannula, snoring, and arterial oxygen saturation using pulse oximetry. Apnea and hypopnea were defined in accordance with standard used criteria. All the recordings were manually scored by the same experienced medical doctor.

Three nonlinear indices (Largest Lyapunov Exponent-LLE, Detrended Fluctuation Analysis-DFA and Approximate Entropy-APEN) were extracted from two respiratory signals (nasal cannula flow-F and thoracic belt movement-T). The oxygen saturation signal (SpO2) from pulse oximetry was also selected. The above signals had a mean duration of 317.5 minutes and were first exported in European Data Format (EDF) to be further processed with the use of signal processing software (Matlab by Mathworks Inc.) in personal computers. The LLE calculation required the use of a command line application by Rosenstein et al as well as a spreadsheet program (Microsoft Excel).

The basic statistical analysis was performed with the use of SPSS for Windows, Version 15.0 (SPSS Inc, Chicago, Illinois). Correlations between the studied or derived parameters were explored with the Pearson's correlation test and differences in the mean observed values between the various OSAHS severity groups were analyzed using the Student's t-test. The statistical significance level was set at p<0.05. The predictive model was created by utilizing the linear regression tool.

ELIGIBILITY:
Inclusion Criteria:

* symptoms compatible with OSAHS
* voluntary participation

Exclusion Criteria:

* presence of dementia
* neuromuscular disorders
* overlap syndrome
* severe cardiac problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Sleep Unit of a tertiary hospital in northern Greece during the years 2005-2008 and who accepted to sign the informed consent form were included in the study. One out of every five consecutive patients was selected in order to ensure randomization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
nonlinear dynamics of respiratory signals | One night
  calculation of nonlinear parameters (DFA, LLE, APEN) from recorded respiratory biosignals (nasal airflow, thoracic movement and SpO2) during sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos K Kaimakamis, MD, MSc, Principal Investigator — Aristotle University Of Thessaloniki; Nikolaos Maglaveras, PhD, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- Sleep Unit of "G. Papanikolaou" General Hospital, Exochi, Greece

REFERENCES:
- [Result] Kaimakamis E, Bratsas C, Sichletidis L, Karvounis C, Maglaveras N. Screening of patients with Obstructive Sleep Apnea Syndrome using C4.5 algorithm based on non linear analysis of respiratory signals during sleep. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:3465-9. doi: 10.1109/IEMBS.2009.5334605. PMID 19964987
- [Derived] Kaimakamis E, Tsara V, Bratsas C, Sichletidis L, Karvounis C, Maglaveras N. Evaluation of a Decision Support System for Obstructive Sleep Apnea with Nonlinear Analysis of Respiratory Signals. PLoS One. 2016 Mar 3;11(3):e0150163. doi: 10.1371/journal.pone.0150163. eCollection 2016. PMID 26937681